CLINICAL TRIAL: NCT06172998
Title: New Perspective on Exploring the Post-apneic Blood Pressure Surge in Patients With Obstructive Sleep Apnea
Brief Title: New Perspective on Exploring the Post-apneic BP Surge in Patients With OSA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu J (Other)
Responsible Party: Sponsor-Investigator, Xu J, professor, Huai'an No.1 People's Hospital
Organization: Huai'an No.1 People's Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Huaian1PH8
Record Dates: First submitted 2023-11-26; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Phentolamine; Nitroglycerin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy subject (No Intervention)
- low BPV group (No Intervention)
- high BPV group (Experimental)
  Interventions: Drug: Phentolamine Injection

INTERVENTIONS:
Drug: Phentolamine Injection — Under patient safety, Phentolamine will be pumped into the OSA patients equipped with PSG and ECG monitoring in a safe dose to prevent sympathetic overactivity. Under patient safety, Nitroglycerin will be pumped into the OSA patients equipped with PSG and ECG monitoring in a safe dose to prevent endothelial dysfunction.
  Other Names: Nitroglycerin
  Arms: high BPV group

SUMMARY:
The nocturnal short-term BPV induced by sleep-breathing events is affected by many factors. The purpose of the study is as follows: (1) to explore the relationship between nocturnal short-term BPV and vascular endothelial function and sympathetic activity in patients with OSA respectively, (2) to explore which play the key role in BP fluctuation, (3) how to prevent the frequent BP fluctuation and arrive at a safe point.

DETAILED DESCRIPTION:
It has been known that nocturnal short-term blood pressure variability (BPV) is a special phenomenon in obstructive sleep apnea (OSA) patients. Nocturnal short-term BPV is a quantitative measure that describes the BP fluctuation over a period of seconds to minutes. It is significantly associated with target organ injury, increased risk of cardio-cerebrovascular events, and increased mortality, independent of mean BP level. Our prior study found that nocturnal BP will temporarily reach the peak during one OSA episode and come to decline rapidly. However, this phenomenon does not occur in all OSA patients. In some severe OSA patients with severe hypoxemia, their BP can still maintain a relatively stable level when one OSA episode. The specific mechanism is still unclear. In physiological conditions, the BP fluctuation caused by each cardiac cycle is affected by vascular function, central sympathetic, arterial reflex, cardiopulmonary reflex, elastic properties of arteries, humoral, and even emotional factors. Therefore, the purpose of the study is as follows: (1) to explore the relationship between nocturnal short-term BPV and vascular endothelial function and sympathetic activity in patients with OSA respectively, (2) to explore which play the key role in BP fluctuation, (3) how to prevent the frequent BP fluctuation and arrive at a safe point.

First, about 300 suspected OSA and 50 healthy subjects under full-night polysomnography (PSG) will be recruited in the sleep medicine center of The Affiliated Huai'an No. 1 People's Hospital of Nanjing Medical University and The First Affiliated Hospital with Nanjing Medical University. All the participants complete the questionnaire which includes clinical medical history, sleep habits, general health, smoking and drinking history, and anthropometric data. When PSG worked, BP was calculated by pulse transit time (PTT) simultaneously and continuously. The electrocardiography data extracted from the entire overnight PSG recordings are visually inspected for accuracy and quality and used for heart rate analysis (HRV) analysis. The next day, 4-5 mL peripheral venous blood samples are obtained from participants in the morning after an overnight fast and used for biochemical analysis. The sympathetic activity could be represented by HRV and Norepinephrine detected by enzyme-linked immunosorbent. Then, brachial artery diameter will be measured after the reactive hyperemia (called flow-mediated dilation, FMD) and nitroglycerin stimulus (called nitroglycerin-mediated dilation, NMD). The FMD and NMD could represent the vascular function. About 80 patients will be in the next plan. On the second day, under patient safety, Phentolamine will be pumped into the OSA patients equipped with PSG and ECG monitoring in a safe dose to prevent sympathetic overactivity. On the third day, under patient safety, Nitroglycerin will be pumped into the OSA patients equipped with PSG and ECG monitoring in a safe dose to prevent endothelial dysfunction. The parameters before and after medicine will be analyzed and compared.

Hypothesis: The investigator predicted that patients who received phentolamine and nitroglycerin injections would lower nocturnal short-term BPV measured by polysomnography

ELIGIBILITY:
Inclusion Criteria:

* medium to severe OSA (apnea-hypopnea index, AHI≥15 events/h) and patients without OSA (AHI<5 events/h)
* age from 18 to 65 years old.

Exclusion Criteria:

* combined with other sleep disorders
* patients with comorbidities, such as hypertension, diabetes, cardiovascular diseases, and cerebrovascular diseases etc
* conditions that potentially affect the accuracy of BPV and endothelial function
* ever-received the treatment of constructive positive airway pressure (CPAP)
* who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with high nocturnal short-term BPV will change | one night

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Xu, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres G, Sanchez-de-la-Torre M, Barbe F. Relationship Between OSA and Hypertension. Chest. 2015 Sep;148(3):824-832. doi: 10.1378/chest.15-0136. PMID 25879807
- [Background] Xu J, Ding N, Zhang X, Wang N, Sun B, Zhang R, Xie X, Wan Z, Gu Y, Zhang S, Hong Y, Huang M, Meng Z. Nocturnal blood pressure fluctuation and associated influential factors in severe obstructive sleep apnea patients with hypertension. Sleep Breath. 2018 Dec;22(4):1045-1052. doi: 10.1007/s11325-018-1634-6. Epub 2018 Mar 9. PMID 29524090
- [Background] Sun B, Ma Q, Shen J, Meng Z, Xu J. Up-to-date advance in the relationship between OSA and stroke: a narrative review. Sleep Breath. 2024 Mar;28(1):53-60. doi: 10.1007/s11325-023-02904-2. Epub 2023 Aug 26. PMID 37632670
- [Background] Xu J, Ding N, Chen L, Zhang Y, Huang M, Wang Y, Meng Z, Zhang X. Inducers of post-apneic blood pressure fluctuation monitored by pulse transfer time measurement in obstructive sleep apnea varied with syndrome severity. Sleep Breath. 2019 Sep;23(3):769-776. doi: 10.1007/s11325-018-1770-z. Epub 2019 Jan 12. PMID 30637570
- [Background] Schutte AE, Kollias A, Stergiou GS. Blood pressure and its variability: classic and novel measurement techniques. Nat Rev Cardiol. 2022 Oct;19(10):643-654. doi: 10.1038/s41569-022-00690-0. Epub 2022 Apr 19. PMID 35440738
- [Background] Sinski M, Lewandowski J, Przybylski J, Bidiuk J, Abramczyk P, Ciarka A, Gaciong Z. Tonic activity of carotid body chemoreceptors contributes to the increased sympathetic drive in essential hypertension. Hypertens Res. 2012 May;35(5):487-91. doi: 10.1038/hr.2011.209. Epub 2011 Dec 8. PMID 22158114
- [Background] Smith RP, Veale D, Pepin JL, Levy PA. Obstructive sleep apnoea and the autonomic nervous system. Sleep Med Rev. 1998 May;2(2):69-92. doi: 10.1016/s1087-0792(98)90001-6. PMID 15310503
- [Background] Narkiewicz K, van de Borne PJ, Montano N, Dyken ME, Phillips BG, Somers VK. Contribution of tonic chemoreflex activation to sympathetic activity and blood pressure in patients with obstructive sleep apnea. Circulation. 1998 Mar 17;97(10):943-5. doi: 10.1161/01.cir.97.10.943. PMID 9529260
- [Background] Narkiewicz K, van de Borne PJ, Pesek CA, Dyken ME, Montano N, Somers VK. Selective potentiation of peripheral chemoreflex sensitivity in obstructive sleep apnea. Circulation. 1999 Mar 9;99(9):1183-9. doi: 10.1161/01.cir.99.9.1183. PMID 10069786
- [Background] Tobaldini E, Costantino G, Solbiati M, Cogliati C, Kara T, Nobili L, Montano N. Sleep, sleep deprivation, autonomic nervous system and cardiovascular diseases. Neurosci Biobehav Rev. 2017 Mar;74(Pt B):321-329. doi: 10.1016/j.neubiorev.2016.07.004. Epub 2016 Jul 7. PMID 27397854
- [Background] Kim YS, Kim SY, Park DY, Wu HW, Hwang GS, Kim HJ. Clinical Implication of Heart Rate Variability in Obstructive Sleep Apnea Syndrome Patients. J Craniofac Surg. 2015 Jul;26(5):1592-5. doi: 10.1097/SCS.0000000000001782. PMID 26114507
- [Background] Pumprla J, Howorka K, Groves D, Chester M, Nolan J. Functional assessment of heart rate variability: physiological basis and practical applications. Int J Cardiol. 2002 Jul;84(1):1-14. doi: 10.1016/s0167-5273(02)00057-8. PMID 12104056
- [Background] Rajendra Acharya U, Paul Joseph K, Kannathal N, Lim CM, Suri JS. Heart rate variability: a review. Med Biol Eng Comput. 2006 Dec;44(12):1031-51. doi: 10.1007/s11517-006-0119-0. Epub 2006 Nov 17. PMID 17111118
- [Background] van der Steen MS, Lenders JW, Graafsma SJ, den Arend J, Thien T. Reproducibility of ambulatory blood pressure monitoring in daily practice. J Hum Hypertens. 1999 May;13(5):303-8. doi: 10.1038/sj.jhh.1000808. PMID 10376847
- [Background] Gesche H, Grosskurth D, Kuchler G, Patzak A. Continuous blood pressure measurement by using the pulse transit time: comparison to a cuff-based method. Eur J Appl Physiol. 2012 Jan;112(1):309-15. doi: 10.1007/s00421-011-1983-3. Epub 2011 May 10. PMID 21556814
- [Background] Ramaekers D, Beckers F, Demeulemeester H, Aubert AE. Cardiovascular autonomic function in conscious rats: a novel approach to facilitate stationary conditions. Ann Noninvasive Electrocardiol. 2002 Oct;7(4):307-18. doi: 10.1111/j.1542-474x.2002.tb00179.x. PMID 12431308
- [Background] Meglic B, Danieli A. Glyceryl trinitrate-induced blood pressure variability decrease during head-up tilt test predicts vasovagal response. Blood Press Monit. 2023 Oct 1;28(5):236-243. doi: 10.1097/MBP.0000000000000653. Epub 2023 Jun 19. PMID 37334541